CLINICAL TRIAL: NCT06553833
Title: Impact of Transfusions and Patient Blood Management on Outcomes in Patients Undergoing Major Surgery
Brief Title: Outcomes of Patient Blood Management in Patients Undergoing Major Surgery
Status: Completed | Type: Observational
Sponsor: Helios Klinik Gotha/Ohrdruf (Other)
Collaborators: HELIOS Hospital, Erfurt, Germany (Other); Matthias Lucas (Unknown)
Responsible Party: Principal Investigator, Petra Seeber, Principal Investigator, Helios Klinik Gotha/Ohrdruf
Other Study IDs: O-PBM3
Record Dates: First submitted 2024-05-05; First posted 2024-08-14 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Major Surgery
Keywords: major surgery; anemia; transfusion; patient blood management
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study group 1: PBM only: Participants in study group 1 receive full PBM while they opted not to receive transfusions.
  Interventions: Other: Patient Blood Management
- Study group 2: PBM with transfusions: Participants in study group 2 receive partial PBM while they opted to receive transfusions. Transfusions are given by physicians encouraged to use a restrictive transfusion strategy. PBM is delivered to participants at a convenient time, resorting to a set of standard PBM measures rather than individualized care.
  Interventions: Biological: Allogeneic transfusion; Other: Patient Blood Management
- Control group: Transfusions only: The control group is treated in an environment where PBM is not implemented and transfusion is the standard therapy for anemia, major bleeding, thrombopenia and coagulopathy beyond the transfusion trigger.
  Interventions: Biological: Allogeneic transfusion

INTERVENTIONS:
Biological: Allogeneic transfusion — Anemia is treated by administering donor red cells, and bleeding or coagulopathy by plasma, platelets or other donor blood products.
  Groups: Control group: Transfusions only; Study group 2: PBM with transfusions
Other: Patient Blood Management — PBM is a strategy to manage the participants own blood. Its focus is on anemia, bleeding and coagulation management (using predominantly pharmaceutical and technological means).
  Groups: Study group 1: PBM only; Study group 2: PBM with transfusions

SUMMARY:
The goal of this observational study is to compare patients who underwent major surgery and who were eligible to receive different management of their red blood count, namely, allogeneic transfusions with or without patient blood management, or blood management alone. Its main questions it aims to answer are:

Which group of patients dies more frequently: Patients who receive patient blood management only, patients who receive patient blood management and transfusions where indicated, or patients who are eligible to receive transfusions only.

Among these groups: which group of patients has more complications during hospital stay? Patients will either receive patients blood management, which is the management of anemia, bleeding and coagulation problems, will receive transfusions, that is, blood from other people, or a mix of both.

DETAILED DESCRIPTION:
Background:

There seems to be a clear relationship between hemoglobin level and inhospital morbidity and mortality. To mitigate negative effects of lower hemoglobin levels, that is, anemia, transfusions are given when the hemoglobin level of the patient reaches a point deemed detrimental by the treating health care personnel. Patient Blood Management (PBM) adds to the armamentarium of anemia therapy, starting typically well before transfusions are given, and sometimes beyond this point. PBM utilizes medical strategies to enhance the patients own red cell mass and to alleviate the ill effects of disease and bleeding on hematopoiesis and hemostasis.

Objective:

The objectives of this study is to investigate the effects of different blood management strategies in patients undergoing major surgery, namely PBM exclusively or PBM with transfusion therapy combined, and compare them to standard transfusion therapy as regards inhospital mortality and morbidity.

Hypothesis:

It is hypothesized that participants who undergo major surgery and who were eligible to receive a combination of PBM and restrictive transfusion regime would have a lower mortality and less complications than participants receiving a liberal transfusion therapy without PBM, while participants opting to receive only PBM without transfusion support will have increased inhospital mortality and morbidity.

Setting:

The study will be performed at HELIOS Klinikum Gotha (HKG) and HELIOS Klinikum Erfurt (HKE) which are two neighboring hospitals with overlapping personnel, purchasing, IT departments and standard operating procedures. Both hospitals offer basic, advanced and specialist care to their communities. HKG offers PBM to their patients, while HKE does not.

Data sources:

Data will be sourced from the hospital information systems of HKG and HKE. Diseases are coded with the ICD-10-GM (International Code of Diseases, Version 10, Germany) and procedures using the OPS code (Procedure Key, analogous to the International Code of Procedures).

Participants:

All adults undergoing major surgery and being treated between June 01, 2008 and December 31, 2020 in HKG and HKE will be eligible for enrollment when they were treated by a specialty that both hospitals offer.

Interventions:

Study group 1: Participants in this group received full PBM measures as clinically appropriate, but were not transfused at all, no matter how low their hemoglobin dropped.

Study group 2:

Participants in this group received convenience measures of PBM and were transfused as deemed necessary in an environment where a restrictive transfusion strategy is encouraged.

Control:

The control group was treated without systematic PBM offered to patients and transfusions were the only standard of care beyond the individual transfusion trigger.

Outcome:

Primary outcome is inhospital mortality. Secondary outcomes are morbidity measures as outlined below.

Study design:

This is a dual-center, retrospective observational cohort study. Reporting of results will be performed in line with the REporting of studies Conducted using Observational Routinely-collected health Data (RECORD) statement extension of the STrengthening the Reporting of Observational studies in Epidemiology (STROBE) statement.

ELIGIBILITY:
Inclusion Criteria:

* adult
* undergoing major surgery

Exclusion Criteria:

* treatment in a non-comparable specialty
* transfer from admitting hospital within 6 h after arrival
* requesting PBM/ transfusion-free therapy but not offered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all hospitalized participants admitted to HELIOS Klinikum Gotha and Erfurt between June 1, 2008 and December 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 25979 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Inhospital Mortality | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Number of dead participants at the end of hospitalization (inhospital mortality)

SECONDARY OUTCOMES:
Local surgical complications | From date of admission to hospital until the date of discharge or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Number of participants with local surgical complications
Acute myocardial infarction | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Number of participants with acute myocardial infarction
Renal injury | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Number of participants with renal injury (according to RIFLE criteria)
Length of stay in hospital | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 1000 months
  Number of days a participant spends in hospital
Readmission | From date of admission to hospital until 30 days thereafter
  Number of participants readmitted to the same hospital within 30 days from first admission
Transfusion reaction | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Number of participants with a documented transfusion reaction
Need of Intensive Care Unit treatment | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Number of participants needing treatment in an Intensive Care Unit
Respiratory complications | From date of admission to hospital until the date of discharge from hospital or date of death from any cause, whichever came first, assessed for the whole hospitalization period, assessed up to 100 months
  Number of participants with respiratory complications, defined as those needing ventilatory assistance

CONTACTS AND LOCATIONS:
Overall Officials: Petra Seeber, Principal Investigator — HELIOS Klinikum Gotha
Locations (1):
- Helios Klinikum, Gotha, Germany

IPD SHARING:
Plan to Share IPD: No